CLINICAL TRIAL: NCT06999564
Title: The Effect of Eft applıed Before Cesarean sectıon on Postpartum feelıngs of Safety, anxıety and postoperatıve paın: RCT
Brief Title: Effects of EFT on Postpartum Safety Perception, Anxiety, and Postoperative Pain After Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Principal Investigator, Hafize Dağ Tüzmen, Asst.Prof., KTO Karatay University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EFT AND CESAREAN SECTION
Record Dates: First submitted 2025-04-13; First posted 2025-05-31 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Pain Management; Anxiety
Keywords: caesarean section; anxiety; sense of course
MeSH Terms: conditions — Agnosia; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This study is a parallel randomized controlled trial on 60 primiparous women with cesarean section pain randomly allocated to EFT and control groups. The study was approved by the Ethics Committee of KTO Karatay University Faculty of Medicine. In addition, the protocol of this study was registered in the Clinical Trials Register. All participants gave written informed consent before data collection. Women were included according to the following criteria: at least primary school graduate, primiparous, planned cesarean section, and postoperative pain of 4 or more according to VAS. Women with chronic diseases such as heart disease, high blood pressure and diabetes, history of miscarriage, placenta previa, mental illness in the past year, use of psychoactive drugs, drug addiction, smoking, and pregnancy complications such as pre-eclampsia, bleeding, intrauterine death and preterm delivery were excluded.
Who Masked: Investigator, Outcomes Assessor
Masking Description: While the pre-tests and post-tests of the study will be administered by a researcher who does not know which groups the participants are assigned to, they will be administered by the lead researcher who is an expert in EFT and the results will be reported by a blind statistician.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EFT (Experimental): Three sessions of face-to-face EFT will be applied to mothers who will have a planned cesarean section three days before delivery. In order to examine the effect of EFT on women's feelings of security, anxiety and pain levels after childbirth, face-to-face EFT will be applied to mothers in the postpartum period after cesarean section.
  Interventions: Behavioral: EFT
- CONTROL (No Intervention): No application was made to the control group. Following the pre-test application, VAS, SUI and STAI-I-SATAI-II post-test data will be applied before and after cesarean delivery. After the data were reported, EFT was applied to the women in the control group individually by the researchers.

INTERVENTIONS:
Behavioral: EFT — EFT involves the following steps:
  1. Identification of the problem that is causing the person distress (e.g., fear of childbirth) and scoring or measuring the severity of this problem.
  2. Tapping with the fingertips on certain points of the face and body, known as correction (i.e., regulation of the energy system), as well as the expression of an emphatic phrase (related to the person's problem and self-acceptance).
  Arms: EFT

SUMMARY:
This study is a parallel randomized controlled trial on 60 primiparous women with cesarean section pain, randomly divided into EFT and control groups. The study was approved by KTO Karatay University Faculty of Medicine Ethics Committee. Women will be included in the study according to the following criteria: at least primary school graduate, primiparous, planned cesarean section and 4 or more postoperative pain according to VAS. Women with chronic diseases such as heart disease, high blood pressure and diabetes, history of miscarriage, placenta previa, mental illness in the past year, psychoactive drug use, drug addiction, smoking, and pregnancy complications such as pre-eclampsia, bleeding, intrauterine death and preterm delivery will be excluded. Data collection will start in June 2025 and will be completed in August 2025.

DETAILED DESCRIPTION:
Caesarean section is a surgical operation used when vaginal delivery is risky for the mother and fetus and can have both long and short-term effects on maternal and infant health. It is known that caesarean sections do not have a proven positive effect on mother-baby health, but may have negative consequences. After cesarean section, women may experience various problems such as inability to perform activities of daily living, breastfeeding problems, inability to actively take care of the newborn, decreased postpartum comfort, anxiety, depression, insomnia and pain.

Postoperative pain, one of the most common complications of cesarean section, plays an important role in ensuring skin-to-skin contact, establishing mother-baby bonding, initiating breastfeeding, the mother's recovery process and maternal-infant health. In addition, women may experience various levels of stress, anxiety and insecurity after cesarean section. Factors such as spousal support, presence of social support resources, attitudes of health personnel, antenatal education about the postpartum period, general well-being of mother and baby, stress, anxiety, depression, mode of delivery, perception of delivery, birth experience, breastfeeding problems, early discharge are factors affecting mothers' sense of security in the postpartum period. Failure to provide a sense of security after birth increases the risk of anxiety and depression in the following periods. Factors that increase anxiety in women after cesarean section include surgical operation, prolonged transition to oral feeding, late mobilization, risk of infection, delayed mother-infant interaction and milk release.

Early detection of post-cesarean anxiety and postpartum sense of security and taking measures to address these conditions can improve the mother's quality of life, reduce anxiety and worry, and contribute to the effective and efficient maintenance of the mother-infant relationship. Reducing postoperative pain is also of great importance in terms of preventing physical complications and chronic pain, relieving depression, improving the quality of life of the individual, providing postpartum comfort and supporting effective breastfeeding. The side effects of pharmacologic methods used to improve postoperative pain and comfort after cesarean section and the inadequacy of these methods have increased the interest in non-pharmacologic approaches. Nonpharmacological techniques include diaphragmatic breathing exercises, Lamaze methods, visualization, meditation, acupuncture, acupressure, reflexology, massage, hypnosis, aromatherapy, prayer therapy, music therapy and EFT. EFT (Emotional Freedom Techniques) envisages pressing and stimulating the meridian crossing points of the organs associated with these emotions in order to improve psychological conditions such as anger, sadness and anxiety. EFT can resolve emotional problems, reduce anxiety levels, make the person feel calmer and think more positively, supporting maternal and fetal health.

A review of the literature shows that mothers have the most problems with pain, breastfeeding and mobilization after cesarean section and need help with these problems; 78% of women who gave birth by cesarean section experience moderate to severe pain, which negatively affects maternal comfort, and mothers who undergo cesarean section experience unbearable pain of different intensities. In the world, anxiety and depression in the postpartum period have increased in the last decade, as Hada et al. (2019) reported in their study. Postpartum depression rates have been reported to be approximately 13% worldwide. Postpartum anxiety and depression are more common in the early postpartum period and in women who gave birth by cesarean section.

EFT has been reported to be effective in many other areas, including the treatment of disorders such as generalized or specific anxiety, morbid fears, depression, posttraumatic stress disorder, chronic pain and addiction. However, so far, no study has examined the effect of EFT on postpartum feelings of safety, anxiety and postoperative pain together. In the light of this information, unlike the studies in the literature, this study will be conducted to examine the effect of EFT applied before cesarean section on postpartum feelings of safety, anxiety and postoperative pain. In this context, anxiety levels, pain intensity and postpartum feelings of safety will be evaluated in the post-cesarean period. Therefore, it is thought that the results obtained from the study will guide future studies and make a significant contribution to the literature.

ELIGIBILITY:
Inclusion Criteria:

* primary school graduate
* primiparous
* planned cesarean section
* Postoperative pain of 4 or more according to VAS.

Exclusion Criteria:

* Heart disease
* high blood pressure
* chronic diseases such as diabetes
* history of miscarriage
* placenta previa
* mental illness in the last year
* use of psychoactive drugs
* drug addiction
* cigarette smoking
* preeclampsia
* bleeding
* intrauterine death
* premature birth

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — will be performed with women who have had a planned caesarean section
Enrollment: 60 (Actual)
Dates: Start 2025-06-02 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-13 (Actual)

PRIMARY OUTCOMES:
EFT for women who had a planned caesarean section | 0-24 hour
  Face-to-face EFT will be applied to mothers in the period after cesarean delivery in order to examine the effect of EFT application between 0-24 hours on womens pain level.
2. EFT for women with a planned cesarean section | 0-24 hour
  Description: By applying EFT face-to-face to mothers in the period after cesarean delivery, the effect of EFT application between 0-24 hours on women's anxiety levels will be examined.

SECONDARY OUTCOMES:
3.EFT for women with a planned cesarean section | 0-24 hour
  EFT for women with a planned cesarean section
  Remove Description: By applying EFT face-to-face to mothers in the period after cesarean delivery, the effect of EFT application between 0-24 hours on women's postpartum confidence levels will be examined.

CONTACTS AND LOCATIONS:
Locations (1):
- Hafize Dağ Tüzmen, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
YES
Supporting Information: Study Protocol
Time Frame: June and was completed in August 2025